CLINICAL TRIAL: NCT04943211
Title: Determination of Molecular Status, as Well as the Efficacy and Safety of Fluorodeoxyglucose (18F-FDG) in PET-CT Imaging in Juvenile Patients With Histiocytosis
Brief Title: Determination of Molecular Status, the Efficacy and Safety of Fluorodeoxyglucose in PET-CT Imaging
Acronym: HISTIOGEN
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Anna Raciborska (Other)
Collaborators: Maria Sklodowska-Curie National Research Institute of Oncology (Other); Łukasiewicz Research Network (Unknown); Wrocław University of Environmental and Life Sciences (Unknown)
Responsible Party: Sponsor-Investigator, Anna Raciborska, Prof Ass, Institute of Mother and Child, Warsaw, Poland
Organization: Institute of Mother and Child, Warsaw, Poland (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: HISTIOGEN.
Record Dates: First submitted 2021-06-21; First posted 2021-06-29 (Actual); Last update posted 2025-04-13 (Actual); Status verified 2025-04

CONDITIONS: Histiocytosis
Keywords: Langerhans cell histiocytosis (LCH); histiocytosis; Positron Emission Tomography (PET); molecular status; paediatric patients
MeSH Terms: conditions — Histiocytosis; Histiocytosis, Langerhans-Cell | interventions — Fluorodeoxyglucose F18

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- R1 low intervention arm (Other): Children of both sexes who meet all inclusion criteria and do not meet any exclusion criteria will be eligible for the study.
  Interventions: Drug: fluorodeoxyglucose (18F-FDG)

INTERVENTIONS:
Drug: fluorodeoxyglucose (18F-FDG) — max 6 MGBq/kg, no more than 100
  Other Names: GLUNEKTIK; SYNEKTIK

SUMMARY:
Prospective, low intervention, open, single-center, non-commercial clinical trial to improve diagnostics in patients with histiocytosis by assessing the molecular profile of the tumor tissues, monitoring its presence in free-circulating DNA, and determining the efficacy of fluorodeoxyglucose (18F-FDG) in PET-CT imaging.

DETAILED DESCRIPTION:
HISTIOGEN clinical study is part of the POLHISTIO project. The POLHISTIO project is a non-commercial clinical trial aimed at optimizing the diagnosis and treatment of juvenile patients with histiocytosis. The project objectives are defined as follows: 1) to estimate the nature and frequency of mutations in patients with histiocytosis in both tumor tissues and free-circulating DNA; 2) to compare molecular test results with clinical data; 3) to evaluate the diagnostic usefulness of the status of molecular analysis (MRD) as a prognostic factor compared with other recognized factors. As part of the HISTIOGEN protocol, an immortalized cell line will be derived to study the pathogenesis of the disease, drug sensitivity, and drug resistance mechanisms. The project is intended to include patients from all over Poland

ELIGIBILITY:
Inclusion Criteria:

1. Patient under 18 years of age at the time of inclusion.
2. Histopathologically confirmed or suspected histiocytosis (based on prior test results).
3. Signing of informed consent for trial participation according with current legal regulations.

Exclusion Criteria:

1. Lack of inclusion criteria.
2. Pregnancy.
3. Other acute or persistent disorders, behaviors or abnormal laboratory test results, which might increase the risk related to the participation in this clinical trial or to taking the study drug, or which might influence the interpretation of the study results, or which, in the investigator's opinion, disqualify a patient from participating in the trial.

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 150 (Estimated)
Dates: Start 2021-04-01 (Actual); Primary Completion 2026-03-30 (Estimated); Study Completion 2026-03-30 (Estimated)

PRIMARY OUTCOMES:
EFS - (event-free survival) | 2 years
  Event-free survival (EFS) was defined as the time interval from the date of diagnosis to the date of disease progression, recurrence, second malignancy, death or to date of last follow-up for patients without events.

SECONDARY OUTCOMES:
OS (Overall Survival) | 2 years
  Overall Survival (OS) was defined as the time interval from the date of diagnosis to the date of death or to last follow-up date.
Molecular relapse (in ct DNA) | 2 years
  Molecular relapse was defined as the time interval from the date of any mutation negativization to the date of positive results of any mutation

CONTACTS AND LOCATIONS:
Overall Officials: Anna Raciborska, Principal Investigator — Mother and Child Institute
Locations (1):
- Mother and Child Institute, Warsaw, Mazovian, Poland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Abla O, Jacobsen E, Picarsic J, Krenova Z, Jaffe R, Emile JF, Durham BH, Braier J, Charlotte F, Donadieu J, Cohen-Aubart F, Rodriguez-Galindo C, Allen C, Whitlock JA, Weitzman S, McClain KL, Haroche J, Diamond EL. Consensus recommendations for the diagnosis and clinical management of Rosai-Dorfman-Destombes disease. Blood. 2018 Jun 28;131(26):2877-2890. doi: 10.1182/blood-2018-03-839753. Epub 2018 May 2. PMID 29720485
- [Background] Andersson D, Fagman H, Dalin MG, Stahlberg A. Circulating cell-free tumor DNA analysis in pediatric cancers. Mol Aspects Med. 2020 Apr;72:100819. doi: 10.1016/j.mam.2019.09.003. Epub 2019 Sep 25. PMID 31563277
- [Background] Badalian-Very G, Vergilio JA, Degar BA, MacConaill LE, Brandner B, Calicchio ML, Kuo FC, Ligon AH, Stevenson KE, Kehoe SM, Garraway LA, Hahn WC, Meyerson M, Fleming MD, Rollins BJ. Recurrent BRAF mutations in Langerhans cell histiocytosis. Blood. 2010 Sep 16;116(11):1919-23. doi: 10.1182/blood-2010-04-279083. Epub 2010 Jun 2. PMID 20519626
- [Background] Donadieu J, Piguet C, Bernard F, Barkaoui M, Ouache M, Bertrand Y, Ibrahim H, Emile JF, Hermine O, Tazi A, Genereau T, Thomas C. A new clinical score for disease activity in Langerhans cell histiocytosis. Pediatr Blood Cancer. 2004 Dec;43(7):770-6. doi: 10.1002/pbc.20160. PMID 15390280
- [Background] Fanti S, Franchi R, Battista G, Monetti N, Canini R. PET and PET-CT. State of the art and future prospects. Radiol Med. 2005 Jul-Aug;110(1-2):1-15. English, Italian. PMID 16163136
- [Background] Goyal G, Heaney ML, Collin M, Cohen-Aubart F, Vaglio A, Durham BH, Hershkovitz-Rokah O, Girschikofsky M, Jacobsen ED, Toyama K, Goodman AM, Hendrie P, Cao XX, Estrada-Veras JI, Shpilberg O, Abdo A, Kurokawa M, Dagna L, McClain KL, Mazor RD, Picarsic J, Janku F, Go RS, Haroche J, Diamond EL. Erdheim-Chester disease: consensus recommendations for evaluation, diagnosis, and treatment in the molecular era. Blood. 2020 May 28;135(22):1929-1945. doi: 10.1182/blood.2019003507. PMID 32187362
- [Background] Haupt R, Minkov M, Astigarraga I, Schafer E, Nanduri V, Jubran R, Egeler RM, Janka G, Micic D, Rodriguez-Galindo C, Van Gool S, Visser J, Weitzman S, Donadieu J; Euro Histio Network. Langerhans cell histiocytosis (LCH): guidelines for diagnosis, clinical work-up, and treatment for patients till the age of 18 years. Pediatr Blood Cancer. 2013 Feb;60(2):175-84. doi: 10.1002/pbc.24367. Epub 2012 Oct 25. PMID 23109216
- [Background] Heitzer E. Circulating Tumor DNA for Modern Cancer Management. Clin Chem. 2019 Oct 31:clinchem.2019.304774. doi: 10.1373/clinchem.2019.304774. Online ahead of print. No abstract available. PMID 31672857
- [Background] Janku F, Diamond EL, Goodman AM, Raghavan VK, Barnes TG, Kato S, Abdel-Wahab O, Durham BH, Meric-Bernstam F, Kurzrock R. Molecular Profiling of Tumor Tissue and Plasma Cell-Free DNA from Patients with Non-Langerhans Cell Histiocytosis. Mol Cancer Ther. 2019 Jun;18(6):1149-1157. doi: 10.1158/1535-7163.MCT-18-1244. Epub 2019 Apr 23. PMID 31015311
- [Background] Murakami I, Gogusev J, Jaubert F, Matsushita M, Hayashi K, Miura I, Tanaka T, Oka T, Yoshino T. Establishment of a Langerhans cell histiocytosis lesion cell line with dermal dendritic cell characteristics. Oncol Rep. 2015 Jan;33(1):171-8. doi: 10.3892/or.2014.3567. Epub 2014 Oct 24. PMID 25351656
- [Background] Raciborska A, Bilska K, Weclawek-Tompol J, Gryniewicz-Kwiatkowska O, Hnatko-Kolacz M, Stefanowicz J, Pieczonka A, Jankowska K, Pierelejewski F, Ociepa T, Sobol-Milejska G, Muszynska-Roslan K, Michon O, Badowska W, Radwanska M, Drabko K. Clinical characteristics and outcome of pediatric patients diagnosed with Langerhans cell histiocytosis in pediatric hematology and oncology centers in Poland. BMC Cancer. 2020 Sep 11;20(1):874. doi: 10.1186/s12885-020-07366-3. PMID 32917181